CLINICAL TRIAL: NCT05866926
Title: A Multicenter, Open-label Extension Study to Investigate the Long-term Safety of FAB122 in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Study to Investigate the Long-term Safety of FAB122 in Patients With Amyotrophic Lateral Sclerosis
Acronym: ADOREXT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: After the analysis of the main ADORE study it is concluded that there is no clinical benefit for the patients.
Sponsor: Ferrer Internacional S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FAB122-CT-2201
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: For ADOREXT study, arms from parent study ADORE have been analyzed.
  Data presented for the FAB122 study group correspond to subjects receiving FAB122 in the ADORE study as well as the ADOREXT study (FAB122-FAB122). Data presented for the placebo study group correspond to subjects receiving placebo in the ADORE study and FAB122 in the ADOREXT study (placebo-FAB122).
Masking Description: All subjects were treated with FAB122 in ADOREXT study, arms from parent study ADORE have been analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAB122 (Experimental): Drug: FAB122 Daily dose 100 mg
  Data presented for the FAB122 study group correspond to subjects receiving FAB122 in the ADORE study as well as the ADOREXT study (FAB122-FAB122).
  Interventions: Drug: FAB122
- Placebo (Experimental): Drug: FAB122 Daily dose 100 mg
  Data presented for the placebo study group correspond to subjects receiving placebo in the ADORE study and FAB122in the ADOREXT study (placebo-FAB122).
  Interventions: Drug: FAB122

INTERVENTIONS:
Drug: FAB122 — FAB122 Daily dose 100 mg

SUMMARY:
A multicenter, open-label extension study to investigate the long-term safety of FAB122 in patients with Amyotrophic Lateral Sclerosis

ELIGIBILITY:
Inclusion Criteria:

1. who completed the full study period in the main ADORE study (FAB122-CT-2001);
2. whom the investigator has no concern and judges tolerable for initiating or continuing treatment with FAB122 from a risk and benefit point of view;
3. a female subject should not be able to become pregnant up to 30 days after the last dose of FAB122 and needs to meet at least one of the following criteria:

   * female who is of reproductive potential and has a negative pregnancy test at baseline and is non-lactating.
   * female subject who is not of reproductive potential is eligible without requiring the use of contraception
4. a male patient must:

   * agree he will not donate sperm during the period he will be using FAB122, AND use a condom during sexual intercourse with pregnant or non-pregnant women of childbearing potential

Exclusion Criteria:

1. Patient who has a medical condition or personal circumstances which, in the opinion of the investigator, will make initiation or continuation of treatment with FAB122 not tolerable for them from a risk and benefit point of view.
2. Patient who discontinued study drug prematurely in the double-blind phase of the study (ADORE Study) for safety reasons.
3. Patient who has received any other investigational drug within the period between last visit of the main study and first visit of the extension study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari de Bellvitge, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Groups:
- FAB122: Drug: FAB122(ADORE)-FAB122(ADOREXT)
  FAB122: FAB122 Daily dose 100 mg Data presented for the FAB122 study group correspond to subjects receiving FAB122 in the ADORE study as well as the ADOREXT study (FAB122-FAB122).
- Placebo: Drug: Placebo(ADORE)-FAB122(ADOREXT)
  FAB122: FAB122 Daily dose 100 mg Data presented for the FAB122 study group correspond to subjects receiving Placebo in the ADORE study and FAB122 in the ADOREXT study (Placebo-FAB122).
Period: Overall Study
Arm/Group | FAB122 | Placebo
Started | 135 | 66
Completed (A subject is considered complete if he/she was ongoing at the time of study early termination.) | 110 | 54
Not Completed | 25 | 12
Not completed — Death | 16 | 9
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Disease progression | 1 | 0
Not completed — other causes | 2 | 1

BASELINE CHARACTERISTICS:
Population: Data presented for the FAB122 study group correspond to subjects receiving FAB122 in the ADORE study as well as in the ADOREXT study (FAB122-FAB122).
  Data presented for the Placebo study group correspond to subjects receiving Placebo in the ADORE study and FAB122 in the ADOREXT study (Placebo-FAB122).
Groups:
- Placebo: Drug: Placebo(ADORE)-FAB122(ADOREXT) FAB122 Daily dose 100 mg Data presented for the Placebo study group correspond to subjects receiving Placebo in the ADORE study and FAB122 in the ADOREXT study (Placebo-FAB122).
- Total: Total of all reporting groups
Arm/Group | FAB122 | Placebo | Total
Number analyzed (Participants) | 135 | 66 | 201
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean (SD) | 58.4 (10.6) | 58.5 (10.5) | 58.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 30 | 87
  Male | 78 | 36 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 28 | 16 | 44
  Not Hispanic or Latino | 94 | 48 | 142
  Unknown or Not Reported | 13 | 2 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 119 | 63 | 182
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 3 | 18
Region of Enrollment [Number; unit: participants]
  Europe | 135 | 66 | 201
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.64 (4.03) | 24.76 (3.23) | 25.35 (3.8)
Weight [Mean (Standard Deviation); unit: KG] | 74.87 (14.83) | 71.07 (13.32) | 73.62 (14.43)
Height [Mean (Standard Deviation); unit: CM] | 170.5 (9.5) | 169 (9.8) | 170 (9.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment Emergent Adverse Events
Description: To evaluate the long-term safety of FAB122 in patients with ALS by assessing Number of Participants experiencing Treatment Emergent Adverse Events, evaluating nature and severity.
  The study duration for these subjects, and therefore the duration of FAB122 treatment, was variable depending on the subject's start date, ranging from 3 to approximately 44 weeks.
Time Frame: approximately 44 weeks
Population: as for baseline characteristics
Measure: Number; unit: Participants
Groups:
- FAB122: Drug: FAB122(ADORE)-FAB122(ADOREXT) FAB122 Daily dose 100 mg
  Data presented for the FAB122 study group correspond to subjects receiving FAB122 in the ADORE study as well as in the ADOREXT study (FAB122-FAB122).
Arm/Group | FAB122 | Placebo
Number analyzed (Participants) | 135 | 66
Participants
  Any TEAE | 77 | 41
  Any Serious AE | 29 | 15
  Any Serious TEAE | 29 | 15
  Any TEAE leading to treatment discontinuation | 7 | 5
  Any AE leading to death | 16 | 9
  TEAE by relationship - Unrelated | 75 | 40
  TEAE by relationship - Related | 6 | 3
  TEAE by Severity - Mild | 52 | 31
  TEAE by Severity - Moderate | 32 | 17
  TEAE by Severity - Severe | 24 | 10

2. Secondary Outcome: The Secondary Efficacy Objective to Evaluate the Effect of Treatment With FAB122 Based on Change From Baseline in ALSFRS-R Until End of Study
Description: Change from baseline in ALSFRS-R total score until the end of the study. Revised Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS-R), Maximum value is 48 points and represents better outcome. Minimum value is 0 and represents worse outcome.
Time Frame: 45 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FAB122: Drug: FAB122(ADORE)-FAB122(ADOREXT) FAB122 Daily dose 100 mg
  Data presented for the FAB122 study group correspond to subjects receiving FAB122 in the ADORE study as well as the ADOREXT study (FAB122-FAB122).
Arm/Group | FAB122 | Placebo
Number analyzed (Participants) | 135 | 66
units on a scale | -4.4 (4.8) | -3.8 (5)

ADVERSE EVENTS:
Time Frame: 45 weeks
Arm/Group | FAB122 | Placebo
All-Cause Mortality (participants affected / at risk) | 16/135 | 9/66
Serious Adverse Events (participants affected / at risk) | 29/135 | 15/66
Other Adverse Events (participants affected / at risk) | 77/135 | 41/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAB122 (N=135) | Placebo (N=66)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (4)
Dysponea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 2 (2) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Lower respiratory track infection (Infections and infestations) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 2 (2)
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 0 (0) | 1 (1)
Hospitalization (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Accute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lypoprotein increased (Investigations) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0)
Apathy (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FAB122 (N=135) | Placebo (N=66)
Urinary track infectious (Infections and infestations) | 11 (14) | 1 (1)
Pneumonia (Infections and infestations) | 6 (7) | 1 (1)
COVID-19 (Infections and infestations) | 4 (4) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Lower respiratory track infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 7 (7) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 5 (6) | 6 (14)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Syncope (Nervous system disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 4 (4) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 3 (3) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Renal Colic (Renal and urinary disorders) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-07-10): https://cdn.clinicaltrials.gov/large-docs/26/NCT05866926/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/26/NCT05866926/SAP_001.pdf